CLINICAL TRIAL: NCT04139421
Title: Effects of Shinrin-Yoku (Forest Bathing) on Psychological Well-being in Urban or Rural Green Space: A Pilot Randomized Controlled Trial
Brief Title: Shinrin-Yoku (Forest Bathing) on Psychological Well-being
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PSY008
Record Dates: First submitted 2019-10-20; First posted 2019-10-25 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Mental Health Wellness
Keywords: Shinrin-Yoku; Forest Bathing; Psychological Well-being; Natural Environment
MeSH Terms: conditions — Psychological Well-Being | interventions — Forest Therapy

STUDY DESIGN:
Intervention Model Description: The randomization will be performed by an independent assessor using a computer-generated list of numbers. Participants in both groups will receive a 3-hour Shinrin-Yoku session in either natural forest or urban green area in Hong Kong.
Who Masked: Participant
Masking Description: Deception will be necessary prior to and during the study to achieve blinding of participants for the prevention of expectation bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urban Green Space group (Active Comparator): This group of participants would experience a 3-hour Shinrin-Yoku session in urban green space.
  Interventions: Behavioral: Shinrin-Yoku
- Rural Green Space group (Experimental): This group of participants would experience a 3-hour Shinrin-Yoku session in rural green space.
  Interventions: Behavioral: Shinrin-Yoku

INTERVENTIONS:
Behavioral: Shinrin-Yoku — Shinrin-Yoku is a traditional Japanese practice of getting in touch with nature through walking in the forest in a relaxed way using all five senses.
  Other Names: Forest Bathing

SUMMARY:
This study will examine the effects of Shinrin-Yoku (forest bathing) as an intervention for enhancing psychological well-being in Chinese population. The main component of Shinrin-Yoku is the use of 5 senses in various activities, which typically includes forest walking, meditation, yoga etc. While Shinrin-Yoku has been widely recognized in Japan as a means of preventative health and stress management, it is still a new concept in some countries. In the existing literature, there is increasing evidence demonstrating the efficacy of Shinrin-Yoku for improving for health promotion. However, there is very limited research examining the effectiveness of Shinrin-Yoku in different types of natural environment and the sustainability of its effects.

DETAILED DESCRIPTION:
This study will be a pilot randomized controlled trial on the effects of Shinrin-Yoku (forest bathing) as an intervention for enhancing psychological well-being in Chinese population. Prior to all study procedures, an online informed consent (with phone support) will be obtained from potential participants. Around 30 eligible participants will be randomly assigned to either the natural forest group or the urban green area group in a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents
* Aged from 18 to 65
* Cantonese language fluency
* a willingness to provide informed consent and comply with the trial protocol.

Exclusion Criteria:

* Pregnant
* Have suicidal ideation
* Using medication or psychotherapy for depression
* Experiencing Depression, Anxiety and Stress
* Having unsafe conditions and are not recommended for physical activity by physicians
* Have major psychiatric, medical or neurocognitive disorders that make participation infeasible based on the research team's judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Profile of Mood States-Short Form | Pre-, post-intervention and 1-month post-intervention
  The POMS-SF is a 30-item scale that measures six different dimensions of mood swings over a period of time. These include: Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment. A five-point scale ranging from "not at all" to "extremely" is administered by experimenters to patients to assess their mood states.

SECONDARY OUTCOMES:
Change in Depression Anxiety Stress Scales-21 | Up to 1 month after the intervention
  DASS-21 is a 21-item scale, comprises of three sub-scales which measures the negative emotional states of depression, anxiety, and stress, over the past week. The DASS is based on a dimensional rather than a categorical conception of psychological disorder, thus it has no direct implications for the allocation of patients to discrete diagnostic categories. However, recommended cutoff scores for conventional severity labels (normal, moderate, severe) are given in the DASS Manual.
Change in Nature-relatedness Scale-6 | Up to 1 month after the intervention
  NR-6 is a 6-item scale assesses the self and experience dimensions of individuals' connection to nature. The NR uses 5-point scale ranging from disagree strongly (1) to agree strongly (5). It is important to respond with the actual feelings rather than how "most people" feel.
Change in Brief Resilience Scale | Up to 1 month after the intervention
  BRS consists of six items, three positively worded items, and three negatively worded items. All six relate to the individual's ability to bounce back from adversity. It was predictably related to personal characteristics, social relations, coping, and health in all samples. The BRS uses 5-point scale ranging from strongly disagree (1) to strongly agree (5).
Change in Insomnia Severity Index | Up to 1 month after the intervention
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Change in Subjective Vitality Scales - State Version | Up to 1 month after the intervention
  SVS is a 7-item scale, comprises of two versions which measures subjective vitality in two level, including individual differences level and state level. The SVS uses 7-point scale ranging from not at all true (1) to very true (7). The state level version assesses the state of subjective vitality rather than its enduring aspect.
Change in Self-Compassion Scale-Short Form | Up to 1 month after the intervention
  SCS-SF is a 12-item scale to evaluates the degree of self-compassion. Ratings on the 5-point Likert scale are obtained on 6 factors, including self-kindness, common humanity, mindfulness, self-judgment, isolation and over-identification. The self-report 13-item SCS-SF explicitly represents the thoughts, emotions, and behaviors associated with self-compassion and includes items that measure how often people respond to feelings of inadequacy or suffering with each of six components.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - The Chinese University of Hong Kong, Hong Kong
  - The Chinese University of Hong Kong, Shatin

IPD SHARING:
Plan to Share IPD: No